CLINICAL TRIAL: NCT06076044
Title: Effects of Transcranial Oscillatory Direct Current Stimulation on the Functions of Cerebral Cortex in Healthy Subjects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Hospital of Hebei Medical University (Other)
Responsible Party: Principal Investigator, Yuan Xing, Attending, Department of Neurology, Principal Investigator, The First Hospital of Hebei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstHebei
Record Dates: First submitted 2023-09-21; First posted 2023-10-10 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Transcranial Direct Current Stimulation; Motor Evoked Potential; Healthy Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy subjects (Experimental): healthy male subjects aged 20-30 years
  Interventions: Device: toDCS 2mA 1Hz; Device: toDCS 2mA 10Hz; Device: tDCS 1mA; Device: sham

INTERVENTIONS:
Device: toDCS 2mA 1Hz — The subgroup treated by transcranial oscillatory direct current stimulation of 2mA and 1Hz.
Device: toDCS 2mA 10Hz — The subgroup treated by transcranial oscillatory direct current stimulation of 2mA and 10Hz.
Device: tDCS 1mA — The subgroup treated by transcranial direct current stimulation of 1mA.
Device: sham — The subgroup treated by sham stimulation.

SUMMARY:
To investigate the effect of transcranial oscillatory direct current stimulation on functions of cerebral cortex (cortical excitability and frequency of eeg) in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male
* Age ranges from 20 to 30 years old
* No history of neurological or psychiatric diseases, no history of chronic illness
* No positive results were found in the examination of the nervous system
* All right-handed according to Edinburgh Handedness Inventory
* The subjects voluntarily participated in this study and signed an informed consent form

Exclusion Criteria:

* Individuals with severe illnesses
* Previous history of brain surgery or epilepsy
* Individuals who experience changes in physical condition during the experiment
* Individuals with metal implants, such as pacemakers, DBS therapists, stents, etc
* Alcoholics

Ages: 20 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The participant eligibility is not based on self-representation of gender identity. The investigators apply the gender eligibility to avoid the influence of female's menstrual cycle.
Enrollment: 15 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
MEP | before treatment and 20, 30, 40, 50, 60 minutes after treatment
  Motor evoked potentials of the right abductor pollicis brevis were collected
Power Spectral Density of EEG | before treatment and right after treatment
  The rest state EEG of the subjects was collected

CONTACTS AND LOCATIONS:
Locations (1):
- the First Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

IPD SHARING:
Plan to Share IPD: No